CLINICAL TRIAL: NCT06191107
Title: Clinical Performance of Removable Partial Dentures With Clasps Made of PEEK
Brief Title: Removable Partial Dentures Made of PEEK
Acronym: KLAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Medical University Innsbruck (Other); Merz Dental GmbH (Unknown)
Responsible Party: Principal Investigator, Thomas Stober, Prof. Dr., University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMA-ID 15379
Record Dates: First submitted 2023-11-28; First posted 2024-01-05 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Tooth Loss
Keywords: Removable Partial Denture; Polyetheretherketone; Oral Health Related Quality of Life
MeSH Terms: conditions — Tooth Loss | interventions — Denture, Partial, Removable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PEEK-RPDs (Experimental): Participants with removable partial dentures made of PEEK
  Interventions: Device: Removable Partial Denture

INTERVENTIONS:
Device: Removable Partial Denture — Integration of removable partial dentures made of PEEK for the treatment of tooth loss.

SUMMARY:
As part of the clinical study, 25 patients each were provided with removable partial dentures with clasps made of PEEK in two centres (University Hospital Heidelberg, Department of Prosthodontics and University Hospital for Dental Prosthetics Innsbruck). The patients were examined over a period of 3 years for the number and type of technical or biological complications and questioned about their oral health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a clasp-anchored removable partial denture

Exclusion Criteria:

* Minors and adults unable to give consent
* Pregnancy or breastfeeding
* Severe general illnesses
* Allergies or other intolerances to one of the materials used (PEEK, PMMA)
* Suspicion of lack of compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Oral-Health-Related Quality of Life | 3 months
  Improvement of Oral-Health-Related Quality of Life (OHRQoL) after incorporation of removable partial dentures made of PEEK (PEEK-RPDs) by using a short version of the validated "Oral Health Impact Profile" questionnaire with 14 questions (OHIP-G 14). A precise evaluation is obtained by adding up the 14 items with their frequency ("never"=0, "hardly"=1, "now and then"=2, "often"=3 and "very often"=4) up to a total value. This value can range from 0 (no limitation of OHRQL) to 56 (severe limitation of OHRQoL). These data are collected before treatment and 3 months after insertion of the PEEK-RPDs.
Biological complications | 3 years
  Biological complications (intolerances, damage to the abutment teeth and/or the periodontium, survival of abutment teeth) after incorporation of PEEK-RPDs. Measurement tool: Study report form. These data are collected half-yearly after insertion of the PEEK-RPDs.
Technical complications | 3 years
  Technical complications (clasp fractures, denture defects) after incorporation of PEEK-RPDs. Measurement tool: Study report form. These data are collected half-yearly after insertion of the PEEK-RPDs.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rammelsberg, Prof. / Head, Study Chair — University Hospital Heidelberg
Locations (1):
- University Hospital Heidelberg, Department of Prosthodontics, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No